CLINICAL TRIAL: NCT00814866
Title: Bone Resorption, Osteoclastogenesis and Adalimumab
Acronym: BROCA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Collaborators: Abbott (Industry)
Responsible Party: Principal Investigator, Artur de Brum-Fernandes, MD, Université de Sherbrooke
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: crcel08045; HUM 07-061
Record Dates: First submitted 2008-12-23; First posted 2008-12-25 (Estimated); Last update posted 2016-10-27 (Estimated); Status verified 2013-12

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid arthritis; arthritis; osteoclasts; bone
MeSH Terms: conditions — Arthritis, Rheumatoid; Arthritis | interventions — Adalimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Adalimumab (Other): Open label
  Interventions: Drug: Adalimumab

INTERVENTIONS:
Drug: Adalimumab — Adalimumab 40 mg sub-cutaneously every two weeks
  Other Names: Humira

SUMMARY:
Osteoclastic bone resorption depends on both the capacity to generate osteoclasts (osteoclastogenesis) and on individual osteoclast activity. The investigators objective is to study the effect of anti-TNF therapy on the number of osteoclast precursors in the peripheral blood of patients with Rheumatoid Arthritis, on in vitro osteoclastogenesis and on osteoclast activity before and during the treatment of patients with Rheumatoid Arthritis with Adalimumab.

DETAILED DESCRIPTION:
Osteoclasts (OCs) are cells specialized in bone degradation that participate in bone and joint destruction in Rheumatoid Arthritis (RA). Experimental models have clearly demonstrated that OCs are essential for local bone resorption in arthritis. In RANKL knockout mice(1; 2), in rats receiving OPG(3-6) or in c-fos(-/-) hTNF transgenic mice(7) induction of arthritis leads to inflammation but not to bone erosion. Systemic osteoporosis is an important comorbidity in RA(8; 9). Increased systemic bone resorption due to OC activation occurs even in early (< 2 years) RA and correlates with disease activity(10). Bisphosphonates are effective in preventing systemic bone loss in inflammatory diseases, but for unknown reasons do not seem to influence periarticular bone erosion and joint destruction. Finally, a systemic factor affecting osteoclastogenesis seems to be present in RA, as shown by an increased formation of OCs from bone marrow of patients with severe arthritis when compared to controls(11).

TNF-alpha is a major pathologic mediator in RA. It may induce bone resorption either directly, stimulating osteoclastogenesis(12; 13) or indirectly, by influencing RANKL, OPG and prostaglandin production by osteoblasts(14; 15). These pathways may be important for the pathophysiology of several diseases such as periodontitis, Rheumatoid arthritis and osteoporosis(16; 17). In mice, TNF-alpha increases the number of osteoclast precursors in vivo but its role may, however, be more complex and implicate also osteoclastogenesis-inhibiting mechanisms(18; 19); in fact, in certain conditions, TNF-alpha may decrease osteoclastogenesis(20), so the in vivo effect of blocking TNF may be difficult to predict from these models.

Anti-TNF agents reduce bone destruction in RA but it is not clear how this effect is achieved since, as described in the preceding paragraph, TNF has been shown to have antagonistic effects in osteoclast formation and activity. Moreover, little is known of the effect of anti-TNF therapy on osteoclast biology in humans.

Working hypothesis

This project is based on two different but closely related hypothesis:

1. Treatment with anti-TNF agents (Adalimumab in this case) may reduce the number of circulating osteoclast precursors, in vitro osteoclastogenesis and in vitro bone resorption.
2. Addition of Adalimumab to the culture medium used to differentiate osteoclasts in vitro may inhibit osteoclastogenesis and bone resorption.

Objectives

Osteoclastic bone resorption depends on both the capacity to generate osteoclasts (osteoclastogenesis) and on individual osteoclast activity. Our objective is to study the effect of anti-TNF therapy on the number of osteoclast precursors in the peripheral blood of patients with RA, on in vitro osteoclastogenesis and on osteoclast activity before and during the treatment of patients with RA with Adalimumab.

Research plan

Trial design : As a clinical trail aimed at studying the impact of anti-TNF treatment on osteoclastogenesis and osteoclast activity we will study one cohort of patients with RA before and at two points after beginning of the therapy, 3 and 6 months, so that each patient will be his/her own control (before/after study). The two time points after introduction of the therapy are needed for two reasons : 1) The time when an eventual effect on the parameters studied may reach its peak is not known and 2) To assure that the parameters measured are stable over time.

Outcomes:

Primary outcomes will be the difference in the following parameters before and after treatment with Adalimumab (3 and 6 months):

1. the number of osteoclast precursor (CD14+) cells in the peripheral blood
2. the number of osteoclasts generated in vitro
3. the amount of bone resorption in vitro

Secondary outcomes:

1. Parallel in vitro differentiation assays (number of osteoclasts generated and amount of bone resorption) in the presence of exogenous Adalimumab in the concentration range found in the plasma of treated patients to detect a direct effect of the medication in vitro in osteoclastogenesis.
2. disease activity defined as a DAS28 score (21; 22)
3. Change in functional status by the M-HAQ (23)

Patient cohort:

Inclusion criteria: Patients satisfying the ACR Criteria for RA(24) and having received a prescription of Adalimumab from a rheumatologist at the Centre hospitalier universitaire de Sherbrooke. Patients having received other anti-TNF therapies are eligible only after 5 half-lives of the previous medication. Patients must be willing to sign an informed consent. Concomitant medication other than anti-TNFs and other biologicals is allowed and the treating rheumatologist can adjust it on the best interest of the patients. This study has, thus, no impact on the routine treatment of the patients. Concomitant medication will be recorded and considered in the final analysis.

Exclusion criteria : Patients under age 18 or not capable or willing to provide informed consent, patients starting Adalimumab less than five half lives after the interruption of a previous anti-TNF therapy.

Sample size and statistics: The sample size was calculated based on the distribution and variance of the primary outcome, i.e. the number of osteoclasts generated in vitro. From a population of 51 normal donors in our laboratory the number of osteoclasts generated was 601.1 ± 156.8 osteoclasts/well (data presented at the 2007 annual meeting of the Canadian Rheumatology Association, in press at the Journal of Rheumatology). We considered a test significance level of 5% (α = 0.05) and the power of 80% to detect a difference of at least 100 osteoclasts/well between the groups (paired two-tailed t-test), which led to a total of 22 patients. Considering a 10% loss due to technical reasons the sample size was established at 25 patients.

Methodology

Blood samples: 50 ml of blood in heparin will be collected from each patient no more than 2 months before the beginning of treatment with Adalimumab and 3 and six months after the first administration of the drug (± 2 weeks). DAS-28, HAQ scores, comorbidities and concomitant medication will be determined and recorded at the same times and the coded data stored in a secure database.

Osteoclast Studies:

Osteoclastogenesis: PBMCs will be isolated from 50 ml of blood by Ficoll-Hypaque gradient and the number of CD14+ OC precursors will be determined by FACS. The whole population of PBMCs will be plated in 48-well tissue culture plates containing a bone slice or a glass slide, and the cells will be allowed to differentiate for 21 days in the presence of recombinant RANKL (75 ng/ml) and M-CSF (10 ng/ml). The cells are then fixed and stained for TRAP activity and with hematoxylin. The number of TRAP+ cells containing three or more nuclei will be counted in each well. Triplicates will be used for each patient. In parallel wells the cells will be incubated in the same conditions but in the presence of Adalimumab in concentration comparable to that found in vivo after treatment.

OC resorptive activity: For bone resorption assays, cells differentiated for 21 days on bone slices will be stained for TRAP and 0.2 % toluidine blue. Resorption surface area will be quantified using the image analysis program, Simple PCI. Parellel assays will be done in the presence of Adalimumab.

Statistical analysis:

The groups before and after intervention will be compared using parametric paired two-tailed tests for the variables with a normal distribution and with non parametric tests whenever appropriate.

Anticipated results

These studies will allow us to determine if treatment with Adalimumab has an effect on the number of circulating osteoclast precursors, on the generation of osteoclasts and on the bone-resorbing activity of these cells. It will also allow to determine if Adalimumab, in concentrations found in vivo, may have a direct impact on human osteoclastogenesis and bone resorption. Perhaps more importantly, correlation of the osteoclast results with the clinical parameters studied may allow us an insight on whether an eventual effect on osteoclasts may correlate with the clinical response to the medication, indicating a possible additional mechanism of action of Adalimumab in Rheumatoid Arthritis.

ELIGIBILITY:
Inclusion Criteria:

* Patients satisfying the ACR criteria for Rheumatoid arthritis and having received a prescription of Adalimumab at the Centre Hospitalier Universitaire de Sherbrooke.

Exclusion Criteria:

* Patients under 18 years old
* Patients unwilling or unable to sign an informed consent
* Patients starting Adalimumab less than five half-lifes after the interruption of a previous anbti-TNF therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2008-09; Primary Completion 2010-09 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
The number of osteoclast precursor (CD14+) cells in the peripheral blood | 0, 3 and 6 months
The number of osteoclasts genereated in vitro | 0, 3 and 6 months
The amount of bone resorption in vitro | 0, 3 and 6 months

SECONDARY OUTCOMES:
Osteoclast differentiation in the presence of exogenous Adalimumab | 0, 3 and 6 months
Disease activity defined by the DAS28 score | 0, 3 and 6 months
Change in functionnal status measured by the M-HAQ | 0, 3 and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Artur Fernandes, MD, PhD, Principal Investigator — Centre de recherche du Centre hospitalier universitaire de Sherbrooke; Gilles Boire, MD, M.Sc., Principal Investigator — Centre de recherche du Centre hospitalier universitaire de Sherbrooke
Locations (1):
- Centre de Recherche Clinique Ethienne Lebel, Fleurimont, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided